CLINICAL TRIAL: NCT02506829
Title: A Randomized Comparative Effectiveness Trial Of Financial Incentives Versus Usual Care For Smokers Hospitalized In The Veterans Affairs Hospital System
Brief Title: Financial Incentives for Smoking Treatment
Acronym: FIESTA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: Robert Wood Johnson Foundation (Other); University of California, Los Angeles (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 72426
Record Dates: First submitted 2015-07-01; First posted 2015-07-23 (Estimated); Last update posted 2020-12-11 (Actual); Status verified 2020-12

CONDITIONS: Smoking; Smoking, Tobacco; Tobacco Use Disorder
Keywords: Inpatients
MeSH Terms: conditions — Smoking; Tobacco Smoking; Tobacco Use Disorder | interventions — Nicotine Replacement Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Usual care (Active Comparator): Usual care in hospital, referral to a smoking cessation Quitline on discharge from hospital.
  Interventions: Behavioral: Smoking cessation counseling (Quitline); Behavioral: Smoking cessation pharmacotherapy (e.g, nicotine replacement therapy)
- Financial Incentives (Experimental): Usual care in hospital, referral to a smoking cessation Quitline on discharge from hospital. Financial incentives for: a) speaking with a coach from the Smoker's Quitline ($50), b) completion of another community-based smoking-cessation program ($50), and/or c) use of pharmacotherapies for smoking cessation at 2 weeks ($50); and d) for smoking cessation, confirmed with the use of a cotinine test at 2 months ($150); and e) for smoking cessation, confirmed with the use of a cotinine test at 6 months after study enrollment ($250).
  Interventions: Behavioral: Smoking cessation counseling (Quitline); Behavioral: Smoking cessation pharmacotherapy (e.g, nicotine replacement therapy); Behavioral: Financial incentives

INTERVENTIONS:
Behavioral: Smoking cessation counseling (Quitline)
Behavioral: Smoking cessation pharmacotherapy (e.g, nicotine replacement therapy)
Behavioral: Financial incentives
  Arms: Financial Incentives

SUMMARY:
The investigators plan to compare the impact of two approaches for smoking cessation on smoking abstinence, use of evidenced-based therapy, and quality of life among a diverse population of patients at the Manhattan campus of the VA New York Harbor Healthcare System, which serves a critical safety-net role for urban veterans. During hospitalization, all smokers will receive usual care. Patients will be randomized to one of two arms: financial incentives plus usual care vs. usual care alone, which includes referral to the state Quitline. All patients enrolled in the study will be offered nicotine replacement therapy. The investigators will conduct follow-up assessments at 2 weeks, 2 months, 6 months and 12 months after discharge. The primary study outcome is smoking abstinence at 6-month follow-up, verified by salivary/urinary cotinine.

ELIGIBILITY:
Inclusion Criteria:

1. age ≥ 18 years,
2. smoked tobacco during the prior 30 days,
3. have an active U.S. phone number and address,
4. can provide consent in English and
5. are in at least the contemplative stage of change for quitting smoking, as assessed by a single measure, readiness to quit

Exclusion Criteria:

1. use only smokeless tobacco,
2. are pregnant or breastfeeding,
3. are discharged to an institution (e.g., nursing home, long-term care facility),
4. are unable to provide informed consent, or do not have cognitive ability to enroll or participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 182 (Actual)
Dates: Start 2015-07 (Actual); Primary Completion 2019-03-05 (Actual); Study Completion 2019-05-20 (Actual)

PRIMARY OUTCOMES:
Smoking abstinence assessed by self-reported and biochemically verified by salivary cotinine | 6 months
  Assessed by self-report questionnaire, and biochemically verified by salivary cotinine

SECONDARY OUTCOMES:
Smoking abstinence assessed by self-report | 6 months
  Assessed by self-report questionnaire
Use of evidence based treatment (e.g. counseling and smoking cessation medications) assessed by discharge prescriptions, Quitline records, receipts, letters and/or self-report | 2 weeks and 2 months
  Assessed by discharge prescriptions, Quitline records, receipts, letters and/or self-report
Quality of life as measured by the EQ5-D and VR-12 | 6 months
  As measured by the EQ5-D and VR-12
Short term return on investment of using financial incentives to promote smoking cessation (Cost analysis) | 12 months
  Cost analysis involving hospital utilization data, electronic health records and patient-reported healthcare utilization
Long term return on investment of using financial incentives to promote smoking cessation (Cost analysis) | 3 years
  Cost analysis involving hospital utilization data, electronic health records and patient-reported healthcare utilization

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Ladapo, MD, PhD, Principal Investigator — University of California, Los Angeles; Scott Sherman, MD, MPH, Principal Investigator — NYU Langone Health
Locations (1):
- New York University School of Medicine, New York, New York, United States

REFERENCES:
- [Derived] French KM, Gonzalez SZ, Sherman SE, Link AR, Malik SZ, Tseng CH, Jumkhawala SA, Tejada B, White A, Ladapo JA. Financial IncEntives for Smoking TreAtment: protocol of the FIESTA trial and FIESTA Oral Microbiome Substudy. Trials. 2018 Nov 21;19(1):646. doi: 10.1186/s13063-018-3003-y. PMID 30463608